CLINICAL TRIAL: NCT02711969
Title: A PhaseⅠStudy of Apatinib Mesylate (YN968D1) 1,000mg in Patients With Unresectable Locally Advanced or Metastatic Gastric Cancer Failed to Standard Therapy
Brief Title: A Study of Apatinib Mesylate (YN968D1) 1,000mg in Gastric Cancer Patient Failed to Standard Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BK-AM-GC102
Record Dates: First submitted 2016-02-26; First posted 2016-03-17 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

ARMS (1):
- Apatinib mesylate (Experimental)
  Interventions: Drug: Apatinib mesylate

INTERVENTIONS:
Drug: Apatinib mesylate — 1,000mg Apatinib mesylate p.o. qd

SUMMARY:
An open study to evaluate the safety of apatinib mesylate (YN968D1) 1,000mg monotherapy in patients with unresectable locally advanced or metastatic Gastric cancer failed to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Subjects with histologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction
* Failure or noncompliance of existing standard treatment without alternative treatment
* Measurable disease measured by proper image examination defined by RECIST 1.1
* Life expectancy ≥ 3 months
* Subject must be suitable for oral administration of study medication
* Subject who can submit a written consent form before participating in the test
* Adequate bone marrow, renal, and liver function
* Electrocorticography(ECOG) performance status ≤ 2
* Ability and willingness to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Pregnant or lactating women
* Therapy with clinically significant systemic anticoagulant or antithrombotic agents within 7 days prior to first scheduled dose of YN968D1
* Hemoptysis within 3 months prior to first scheduled dose of YN968D1
* Cytotoxic chemotherapy, immunotherapy, radiotherapy or other targeted therapies within 4 weeks (6 weeks in cases of mitomycin C, nitrosourea, lomustine) prior to first scheduled dose of YN968D1
* Surgery or biopsy within 28 days prior to first scheduled dose of YN968D1
* Minor surgery within 7 days prior to first scheduled dose of YN968D1
* Patients who have experience using YN968D1 before
* Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9 and CYP2C19
* Known history of human immunodeficiency virus infection (HIV)
* Medical history of other cancers (including blood cancer) in the 5 years
* Radiology therapy to target lesion within 28 days, or diagnosis of other cancer within 14 days prior to first scheduled dose of YN968D1
* History of bleeding diathesis or bleeding within 14 days prior to enrollment
* Medical history of clinically significant thrombosis (bleeding or clotting disorder) within the past 3-months
* History of non-malignant GI bleeding, gastric stress ulcerations, or peptic ulcer disease within the past 3-months
* History of idiopathic or hereditary angioedema, sickle cell or any hemolytic anemia
* History of uncontrolled hypertension that in the opinion of the investigator
* Complete Left bundle branch block (LBBB) or bifascicular (RBBB and left anterior or posterior hemi-block)
* Clinically significant S-T segment or T wave abnormality
* Abnormal atrial fibrillation
* History of ECOG or left ventricular ejection fraction (LVEF) abnormality during last 3 months in the opinion of the investigator
* Myocardial infarction or unstable angina pectoris within 6 months prior to starting study medication
* Congestive heart failure (New York Heart Association class III-IV)
* History of other significant cardiovascular disease or vascular disease within the last 6 months
* History of clinically significant glomerulonephritis, biopsy proven tubulointerstitial nephritis, crystal nephropathy, or other renal insufficiencies Treatment with an investigational agent within the longest time frame of either 5 half-lives or 30 days of initiating study drug
* Half-life of other investigator drug is not passed over fivefold or 30 days prior to clinical trial
* Known recreational substance use or psychiatric illness that, in the opinion of the Investigator, may affect compliance with scheduled visits
* Known hypersensitivity to YN968D1 or components of the formulation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) of Apatinib mesylate in patients with unresectable locally advanced or metastatic gastric cancer | First 28 days of dosing
  Graded and described using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.03

SECONDARY OUTCOMES:
Incidence of Adverse events (AEs), Serious AEs (SAEs), clinical laboratory abnormalities, and ECG abnormalities | From date of registration to time of first progressive disease(PD) or death, an average of 1 year
  Incidence and severity of treatment-related adverse events reported and their relationship to Apatinib mesylate will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.3)
Duration of Response(Stable disease, partial response or Complete response) | From date of registration to time of first progressive disease(PD) or death, an average of 1 year
  Tumor response and progression will be evaluated using RECIST v 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, PhD, Principal Investigator — Seoul Asan Medical Center
Locations (1):
- Asan medical center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Derived] Kang YK, Ryu MH, Hong YS, Choi CM, Kim TW, Ryoo BY, Kim JE, Weis JR, Kingsford R, Park CH, Jang S, McGinn A, Werner TL, Sharma S. Phase 1/2a Study of Rivoceranib, a Selective VEGFR-2 Angiogenesis Inhibitor, in Patients with Advanced Solid Tumors. Cancer Res Treat. 2024 Jul;56(3):743-750. doi: 10.4143/crt.2023.980. Epub 2024 Jan 18. PMID 38271925